CLINICAL TRIAL: NCT07213882
Title: A Phase 1, Multicenter, Open-label, Prospective, First-in-human Dose-escalation Clinical Trial of Domain Therapeutics' Anti-CCR8 Monoclonal Antibody (DT-7012) in Patients With Relapsed or Refractory Cutaneous T-cell Lymphomas (CTCL)
Acronym: CITY
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Domain Therapeutics SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP240605
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Cutaneous T Cell Lymphoma (CTCL); Mycosis Fungoides; Sezary Syndrome
Keywords: Cutaneous T Cell Lymphoma; Mycosis Fungoides; Sezary Syndrome
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome

STUDY DESIGN:
Intervention Model Description: Single arm, open-label, multicenter prospective phase 1 dose-escalation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single agent DT-7012 (Experimental)
  Interventions: Drug: DT-7012

INTERVENTIONS:
Drug: DT-7012 — This study use the Bayesian one-stage time-to-event continual reassessment method (TITE-CRM) design for dose finding phase I clinical trials, using an empirical dose-toxicity model with linear weights. A maximum total of 30 patients with CTCL, given 4 candidate dose levels (0.3; 1.0; 3.0; 10.0 mg/kg) will be dose-assigned starting from 1mg/kg dose level, in cohorts of 1 patient and including safety rules notably to ensure staggered accrual.

SUMMARY:
Cutaneous T-cell lymphomas (CTCL) are a heterogeneous group of lymphomas characterized by a primary involvement of the skin. Among them, mycosis fungoides (MF) and Sézary syndrome (SS) are the most common subtypes. SS is defined as erythroderma (erythema of the entire skin surface), and circulating tumor blood cells. The circulating tumor T cells express CD4 and may lose expression of CD7 and CD26, while exhibiting in most cases aberrant expression of CD158k (KIR3DL2), which is a surface marker of Sézary cells. CCR8 is a surface marker of tumor-infiltrating regulatory T cells. It has recently be observed that CCR8 was expressed by tumor cells in CTCL and other peripheral T-cell lymphomas. CCR8 is expressed by skin resident-memory T cells which are believed to be the tumor cell-of-origin in mycosis fungoides. Domain Therapeutics (DT) showed the in vitro efficacy of their proprietary anti-CCR8 mAb DT7012 in the depletion of CTCL cells. Therapeutic depletion of CCR8-expressing cells by DT-7012 could eliminate tumor cells and activate the anti-tumor immunity in CTCL. We hypothesize that treatment with DT-7012 is effective in the treatment of relapsed or refractory (R/R) CTCL as advanced MF and SS.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Patients (≥18 years) with no upper age limit
2. Confirmed diagnosis of mycosis fungoides or Sezary syndrome
3. Stage IB to IVB in the ISCL / EORTC classification
4. Relapsed or refractory (no response) after at least two systemic treatments
5. ECOG performance status 0-1
6. Adequate liver function:

   * Total bilirubin ≤ 1.5 xULN, or Direct bilirubin ≤ 1.5xULN if total bilirubin is >1.5xULN, or total bilirubin >1.5 xULN if elevated total bilirubin is attributed to Gilbert's syndrome or to histologically-proven liver involvement by CTCL
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2,5 x ULN, unless elevated to up to 5 x ULN due to CTCL
7. Adequate hematological function:

   * Absolute neutrophil count of ≥ 1.5 G/L without G-CSF support for at least 7 days
   * Platelet count of ≥ 75 G/L without platelet transfusion within 7 days
   * Hemoglobin ≥ 9 g/dL without RBC transfusion within 7 days
8. Adequate renal function: creatinine clearance calculated by Cockcroft & Gault formula of ≥ 50 mL/min
9. HBV: negative blood HBs Ag or blood HBV DNA. Vaccinated patients may be included. Patients with HBc antibody may be included if HBV DNA is negative
10. HCV: negative HCV serology, or negative HCV RNA if HCV serology is positive
11. HIV: negative HIV serology
12. Negative serum or urinary pregnancy test within 7 days or at baseline prior to study treatment in women of childbearing potential
13. Patients must agree to use a highly effective contraceptive method from inclusion until:

    * If the patient is a male: at least 6 months after the last dose of DT-7012. Men must refrain from donating sperm during this same period
    * If patient is a female of childbearing potential: at least 6 months after the last dose of DT-7012
14. Patients must have the following minimum wash-out from previous treatments:

    * 12 weeks for total skin electron beam irradiation,
    * 4 weeks for monoclonal antibodies
    * 3 weeks for local radiation therapy, systemic cytotoxic anticancer therapy, treatment with other anti-neoplastic investigational agents
    * 3 weeks for systemic retinoids, interferons, vorinostat, romidepsin, fusion proteins
    * 3 weeks for phototherapy
    * 2 weeks for topical therapy (including steroids, retinoids, nitrogen mustard or imiquimod). Topical steroids and oral steroids (10 mg prednisone equivalent/day maximum) are allowed, if the patient has been on a stable dose with stable symptoms for at least 4 weeks prior to study entry.
15. Patient covered by any social security system (registered or being a beneficiary of such a scheme) for French participants only
16. Signed informed consent

Exclusion Criteria:

1. Known central nervous system involvement by CTCL
2. Participation in any study of a health product within 30 days prior to study entry
3. Patients with a history of other malignancies during the past three years (except for: non-melanoma skin cancer, lymphomatoid papulosis, curatively treated localized prostate cancer, curatively treated localized breast cancer, resected thyroid cancer, biopsy proven cervical intraepithelial neoplasia or cervical carcinoma in situ, which are not considered exclusion criteria).
4. Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), or angina, myocardial infarction, cerebrovascular accident, transient ischemic attack within 6 months prior to study entry
5. Any severe acute or chronic medical or psychiatric condition
6. Patients with immunodeficiency
7. Any active systemic viral, bacterial, or fungal infection requiring systemic antibiotics within 1 week prior to first study drug dose
8. Chronic use of systemic corticosteroids of prednisone or equivalent >10 mg prednisone equivalent/day for a chronic condition (washout of 8 days from start of treatment is accepted)
9. Other immunosuppressive therapies are also excluded, (washout of 7 days from start of treatment is accepted)
10. Autologous Hematopoietic Stem Cell Transplantation (HSCT) within 100 days prior to DT-7012 infusion
11. Prior allogeneic HSCT
12. Prior solid organ transplantation
13. Patient with history of confirmed progressive multifocal leukoencephalopathy
14. Known or suspected allergies, hypersensitivity, or intolerance to DT-7012 or its excipients
15. Pregnant or breast-feeding woman, or desire (for both man and woman participant) to conceive a child within 6 months after end of treatment
16. Patient under guardianship or curatorship and protected adults or unable to consent
17. Coagulation disorder contra indicating intravenous infusion
18. History of anaphylactic reaction following vaccination or immunotherapy
19. History or current immune pneumonitis or interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) defined by any treatment-emergent adverse event (TEAE) not attributable to the disease or disease-related processes | Up to 12 months
  Any Grade ≥ 3 non-hematologic toxicity lasting at least 7 days is considered
  DLT, EXCEPT for:
  * Isolated laboratory findings with no clinical signs or symptoms,
  * Grade 3 fatigue, nausea, vomiting, diarrhea, or other manageable constitutional symptom that is responsive to supportive therapy and resolves to Grade ≤ 2 (or baseline if baseline is Grade ≥ 2) within 72 hours
  Any Grade ≥ 3 hematologic toxicity is considered DLT, EXCEPT for:
  * Grade 3 neutropenia (without fever and not requiring growth factor support) lasting for less than 7 days,
  * Grade 3 thrombocytopenia without clinically significant bleeding or requiring platelet transfusion,
  * Grade 3 leukopenia/lymphopenia,
  * Grade 3 anemia that does not require transfusion.

SECONDARY OUTCOMES:
Incidence of Adverse events | Up to 12 months
  Adverse Events (AEs), Serious Adverse Events (SAEs), Drug related AEs, Drug related SAEs, Adverse Events of Special Interest (AESI)
Objective Response Rate | At 3 months
Complete Response (CR) | At 3 months
Partial Response (PR) | At 3 months
Maximum concentration (Cmax) of DT-7012 | Up to 12 months
  At each administration
Trough concentration (Cmin) of DT-7012 | Up to 12 months
  At each administration
Area under the curve (AUC₀-₇) for the first administration | Up to 12 months
  from time 0 to day 7
Area under the curve (AUC₀-₇) for the fourth administration | Up to 12 months
  from time 0 to day 7
Accumulation index (AI) | Up to 12 months
  Expressed as the ratio of concentrations between the fourth and first administration
Accumulation index (AI) | Up to 12 months
  Expressed as the ratio of AUC between the fourth and first administration
Presence of anti-drug antibodies | Up to 12 months
Presence of pruritus | At 3 months
  Assessed by a visual analogue scale (VAS)
Presence of pruritus | At 6 months
  Assessed by a visual analogue scale (VAS)
Presence of pruritus | At 12 months
  Assessed by a visual analogue scale (VAS)
Health Related Quality of Life | At 3 months
  By a standardized skin-specific questionnaire (SkinDex29). Total score varies from 0 to 100. The higher the score the lower the quality of life
Health Related Quality of Life | At 6 months
  By a standardized skin-specific questionnaire (SkinDex29). Total score varies from 0 to 100. The higher the score the lower the quality of life
Health Related Quality of Life | At 12 months
  By a standardized skin-specific questionnaire (SkinDex29). Total score varies from 0 to 100. The higher the score the lower the quality of life
Health Related Quality of Life | At 3 months
  By the EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30). Total score varies from 0 to 100. The higher the score the lower the quality of life.
Health Related Quality of Life | At 6 months
  By the EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30). Total score varies from 0 to 100. The higher the score the lower the quality of life.
Health Related Quality of Life | At 12 months
  By the EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30). Total score varies from 0 to 100. The higher the score the lower the quality of life.
Time to next treatment (TTNT) | Up to 12 months
  Time from initiation of DT-7012 until the time of initiation of any systemic treatment or total-skin treatment (phototherapy or TSEB).
Disease control rate | At 3 months
  Defined as complete, partial response or stable disease
Disease control rate | At 6 months
  Defined as complete, partial response or stable disease
Disease control rate | At 12 months
  Defined as complete, partial response or stable disease
Duration of response (DoR) | Up to 12 months
  Time from measurement of CR/PR (whichever is first recorded) until the date of documented recurrent or progressive disease, assessed in responder patients only
Progression-Free-Survival | Up to 12 months
  Defined with the time from the first DT-7012 administration to progressive disease, relapse, death, or last follow-up.

OTHER OUTCOMES:
Percentage of of positive cells within the infiltrate by immunohistochemistry | At baseline
  Expression of CCR8, on tumor and reactive cells, in skin and blood
Percentage of of positive cells within the infiltrate by immunohistochemistry | At 3 months
  Expression of CCR8, on tumor and reactive cells, in skin and blood
CCR8 mean fluorescence intensity by flow cytometry in peripheral blood | At baseline
CCR8 mean fluorescence intensity by flow cytometry in peripheral blood | At 1 month
CCR8 mean fluorescence intensity by flow cytometry in peripheral blood | At 3 months
Percentage of cells positive | At baseline
  Exhaustion markers PD1, TIGIT, Tregs markers CD25 and FoxP3, activation markers CD69, CD25 and cell markers - CD68, CD163 macrophages, CD8 T cells) will be studied by flow cytometry in peripheral blood
Percentage of cells positive | At 1 month
  Exhaustion markers PD1, TIGIT, Tregs markers CD25 and FoxP3, activation markers CD69, CD25 and cell markers - CD68, CD163 macrophages, CD8 T cells) will be studied by flow cytometry in peripheral blood
Percentage of cells positive | At 3 months
  Exhaustion markers PD1, TIGIT, Tregs markers CD25 and FoxP3, activation markers CD69, CD25 and cell markers - CD68, CD163 macrophages, CD8 T cells) will be studied by flow cytometry in peripheral blood
Percentage of CCR8-positive tumor T cells and Tregs | At baseline
  By multiplex Immunofluorescence in skin
Percentage of CCR8-positive tumor T cells and Tregs | At 3 months
  By multiplex Immunofluorescence in skin
Percentage of the blood tumor clone in skin and blood (in both cellular and cell-free DNA) | At baseline
Percentage of the blood tumor clone in skin and blood (in both cellular and cell-free DNA) | At 3 months

IPD SHARING:
Plan to Share IPD: Undecided